CLINICAL TRIAL: NCT02555085
Title: Phase 1 Randomized, Blinded, Placebo-Controlled Study of Single Ascending Doses of BIIB063 in Healthy Volunteers
Brief Title: Single Ascending Doses of BIIB063 in Healthy Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Clinical study terminated due to preclinical safety findings in non-human primates.
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 234HV101; 2015-001283-18 (EudraCT Number)
Record Dates: First submitted 2015-08-27; First posted 2015-09-21 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- IV Dose 1 (Experimental): Single ascending IV dose or matching placebo based on body weight recorded on Day 1
  Interventions: Biological: BIIB063; Other: Placebo
- IV Dose 2 (Experimental): Single ascending IV dose or matching placebo based on body weight recorded on Day 1
  Interventions: Biological: BIIB063; Other: Placebo
- IV Dose 3 (Experimental): Single ascending IV dose or matching placebo based on body weight recorded on Day 1
  Interventions: Biological: BIIB063; Other: Placebo
- IV Dose 4 (Experimental): Single ascending IV dose or matching placebo based on body weight recorded on Day 1
  Interventions: Biological: BIIB063; Other: Placebo
- IV Dose 5 (Experimental): Single ascending IV dose or matching placebo based on body weight recorded on Day 1
  Interventions: Biological: BIIB063; Other: Placebo
- IV Dose 6 (Experimental): Single ascending IV dose or matching placebo based on body weight recorded on Day 1
  Interventions: Biological: BIIB063; Other: Placebo
- IV Dose 7 (Experimental): Single ascending IV dose or matching placebo based on body weight recorded on Day 1
  Interventions: Biological: BIIB063; Other: Placebo
- SC Dose (Experimental): Single SC dose or matching placebo
  Interventions: Biological: BIIB063; Other: Placebo

INTERVENTIONS:
Biological: BIIB063 — Single ascending IV dose
Other: Placebo — Single dose

SUMMARY:
The primary objective of the study is to evaluate the safety and tolerability of single ascending intravenous (IV) doses and a single subcutaneous (SC) dose of BIIB063 in healthy volunteers. The secondary objectives of the study are to estimate the PK parameters of single ascending IV doses of BIIB063; to estimate the PK parameters and absolute bioavailability (F) of a single SC dose of BIIB063; and to evaluate the immunogenicity of single ascending doses of BIIB063.

ELIGIBILITY:
Key Inclusion Criteria:

* All male subjects and all female subjects of childbearing potential must practice at least 1 highly effective method of contraception (i.e., contraceptive measure with a failure rate of <1% per year; estrogen-containing contraceptives are prohibited) during the study and be willing and able to continue contraception for 4 months after being dosed with study treatment. Male subjects must also be willing to refrain from sperm donation for at least 4 months after the last dose of study treatment. Male subjects must not have unprotected sexual intercourse with a female who is pregnant or breastfeeding during the study.
* Must have a body mass index between 18 and 30 kg/m2, inclusive.
* Must be in good health as determined by the Investigator, based on medical history, physical examination, and 12-lead ECG.

Key Exclusion Criteria:

* History of or positive test result at screening for human immunodeficiency virus, hepatitis C virus antibody, or hepatitis B virus (defined as positive for hepatitis B surface antigen [HBsAg] or hepatitis B core antibody [HBcAb]).
* History of any clinically significant cardiac, endocrine, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, or other major disease, as determined by the Investigator.
* Personal or family history of cardiovascular disease under the age of 50 years, inherited disorder of coagulation (e.g., Factor V Leiden, protein C or S deficiency), or anti-phospholipid Ab syndrome (APS).
* History of meningococcal vaccination or meningococcal meningitis, or history of hypersensitivity to single components of meningococcal vaccines (including MENVEO), any other CRM197, diphtheria toxoid, or meningococcal-containing vaccine.
* History of tuberculosis (TB) or positive QuantiFERON®-TB Gold test
* Personal history of thromboembolic events
* Treatment with any prescription or over-the-counter medication within 14 days prior to randomization (excluding vitamins, dietary supplements, herbal preparations, progestin-only birth control, and paracetamol up to 4 g/day for no more than 5 consecutive days).
* Current enrollment or a plan to enroll in any interventional clinical study in which an investigational treatment or approved therapy for investigational use is administered within 3 months
* Current enrollment or a plan to enroll in any other drug, biologic or device clinical study, or treatment with an investigational drug or approved therapy for investigational use within 3 months
* Blood donation (1 unit or more) within 3 months prior to randomization.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2015-09-30 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2016-06-01 (Actual)

PRIMARY OUTCOMES:
Number of participants experiencing Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to week 12
Number of participants with clinically significant laboratory assessment abnormalities | Up to week 12
Number of participants with clinically significant Vital sign abnormalities | Up to week 12
Number of participants with clinically significant 12-lead electrocardiograms (ECGs) abnormalities | Up to week 12
Number of participants with clinically significant physical examination abnormalities | Up to week 12
Change in antibody titers of vaccine immunization for tetanus | Up to week 12
Change in antibody titers of vaccine immunization for diphtheria | Up to week 12
Change in antibody titers of vaccine immunization for pneumococcus | Up to week 12

SECONDARY OUTCOMES:
PK parameter of single-ascending IV doses of BIIB063: Area under the concentration-time curve from time zero to the time of the last measurable sample (AUClast) | Up to week 12
PK parameter of single-ascending IV doses of BIIB063: Area under the concentration-time curve from time zero to infinity (AUCinf) | Up to week 12
PK parameter of single-ascending IV doses of BIIB063: Maximum observed concentration (Cmax) | Up to week 12
PK parameter of single-ascending IV doses of BIIB063: Time to reach maximum observed concentration (Tmax) | Up to week 12
PK parameter of single-ascending IV doses of BIIB063: Terminal elimination half-life (t1/2) | Up to week 12
PK parameter of single-ascending IV doses of BIIB063: Clearance (CL) | Up to week 12
PK parameter of single-ascending IV doses of BIIB063: Volume of distribution at steady state (Vss) | Up to week 12
PK parameter of a single SC dose of BIIB063: Area under the concentration-time curve from time zero to the time of the last measurable sample (AUClast) | Up to week 12
PK parameter of a single SC dose of BIIB063: Area under the concentration-time curve from time zero to infinity (AUCinf) | Up to week 12
PK parameter of a single SC dose of BIIB063: Maximum observed concentration (Cmax) | Up to week 12
PK parameter of a single SC dose of BIIB063: Time to reach maximum observed concentration (Tmax) | Up to week 12
PK parameter of a single SC dose of BIIB063: Terminal elimination half-life (t1/2) | Up to week 12
PK parameter of a single SC dose of BIIB063 Apparent total body clearance (CL/F) | Up to week 12
PK parameter of a single SC dose of BIIB063: Apparent volume of distribution during terminal elimination phase (Vz/F) | Up to week 12
PK parameter of a single SC dose of BIIB063: Absolute Bioavailability (F) | Up to week 12
Number of participants with positive serum anti-BIIB063 antibodies | Up to week 12
Percentage of participants with positive anti-BIIB063 titers within 12 weeks after administration of BIIB063 | Up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Research Site, Leeds, West Yorkshire, United Kingdom